CLINICAL TRIAL: NCT06347445
Title: Turkish Nationwide SurvEy of Glycemic and Other Metabolic Parameters of Patients With Diabetes Mellitus-2 (TEMD-2 Study)
Acronym: TEMD-2
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, cem haymana, Associate Proffesor, Gulhane School of Medicine
Other Study IDs: GSM012024
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus
Keywords: glycemic regulation; metabolic control; sleep disorder; sexual dysfunction; depression
MeSH Terms: conditions — Diabetes Mellitus; Sleep Wake Disorders; Sexual Dysfunction, Physiological; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diabetes mellitus: Patients with type 1 or type 2 diabetes who were under follow-up in the same center for at least a year.
  Interventions: Other: There is no intervention.

INTERVENTIONS:
Other: There is no intervention. — There is no intervention.

SUMMARY:
This study evaluates the metabolic control status, cardiovascular risk and frequency of comorbidities in diabetic patients followed in tertiary treatment centers in Turkey.

DETAILED DESCRIPTION:
Diabetes mellitus is one of the most common chronic diseases worldwide.The prevalence of diabetes is increased significantly in Türkiye, from 7.2 % in 2002 to 13.7% in 2012. This increasing prevalence leads to serious public health problems and a significant economic burden. Many important diseases such as hypertension and dyslipidemia accompany the picture in diabetic patients. The optimal treatment of diabetes and prevention of diabetic complications, especially the cardiovascular outcomes, is utmost important. Although achieving glycemic targets in patients with diabetes is of great importance, blood glucose is not the only predictor of cardiovascular outcome in diabetes. Optimization of other metabolic parameters such as lipids, arterial blood pressure (ABP), and body weight as well as a healthy lifestyle are utmost important.

Common problems in diabetic patients, such as sleep disorders and sexual dysfunction, affect glycemia regulation in these patients.There is little data on the frequency of these diseases in diabetic patients in Türkiye.

In the TEMD-1 study conducted in 2017, the rates of diabetic patients achieving metabolic goals and the factors affecting these rates were revealed in Turkish patients with diabetes. The findings obtained in the current study will be compared with the findings in 2017, and in addition, the frequency of comorbidities such as sleep disorder, sexual dysfunction, and depression will be tried to be revealed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or type 2 diabetes
* Upper than 18 years old
* To be under follow-up in the same center for at least one year.

Exclusion Criteria:

* Pregnant or lactation period
* Younger than 18 years old
* History of psychiatric disorders interfering cognition or compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 or type 2 diabetes who were under follow-up in the same tertiary endocrine unit for at least a year were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 5707 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Glycemia control status of Turkish adult patients with diabetes mellitus | 7 days
  Glycemia control will be defined as good control if the mean HbA1c level of patients < 7% or poor control if the mean HbA1c level of patient between 7% and 9% and very poor control if the mean HbA1c level of patient > 9%
Blood pressure control status of Turkish adult patients with diabetes mellitus | 7 days
  Home blood pressure <135/85 mmHg or office blood pressure <140/90 mmHg will be defined as under control.
Lipid control status of Turkish adult patients with diabetes mellitus. | 7 days
  Triglyceride < 150 mg/dl, LDL-C <55 mg/dl, <70 mg/dl and < 100 mg/dl according to the cardiovascular risk status, HDL-C > 40 mg/dl for men, and HDL-C > 50 mg/dl for women will be defined as under control.
Weight control status of Turkish adult patients with diabetes mellitus. | 7 days
  Body mass index < 30 kg/m2 will be defined as under control. Weight and height will be combined to report body mass index in kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Sonmez, Prof., Principal Investigator — Ankara Guven Hospital
Locations (1):
- Gulhane School of Medicine Department of Endocrinology and Metabolism, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No